CLINICAL TRIAL: NCT05025813
Title: A Phase 2 Study of De-escalation in Resectable, Locally Advanced Cutaneous Squamous Cell Carcinoma With the Use of Neoadjuvant Pembrolizumab - DESQUAMATE
Brief Title: Neoadjuvant Pembrolizumab in Cutaneous Squamous Cell Carcinoma
Acronym: DESQUAMATE
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Queensland Health (Other Government)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Dr Rahul Ladwa, Medical Oncologist, PAH, Queensland Health
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Ladwa59935
Record Dates: First submitted 2021-06-14; First posted 2021-08-27 (Actual); Last update posted 2022-08-01 (Actual); Status verified 2022-07

CONDITIONS: Cutaneous Squamous Cell Carcinoma of the Head and Neck; Head and Neck Cancer
Keywords: Pembrolizumab; Immunotherapy; Radiation Therapy; Radiotherapy; Neoadjuvant; Radical Neck Dissection
MeSH Terms: conditions — Head and Neck Neoplasms | interventions — pembrolizumab; Neck Dissection

STUDY DESIGN:
Intervention Model Description: Multi-centre, open-labelled, non-randomised, single-arm phase 2 study of Pembrolizumab in participants aged 18 years or older with locally advanced (LA) Stage II-IV resectable cSCC.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Arm A (Experimental): Neoadjuvant Pembrolizumab 4 cycles, 200mg IV Q3W followed by interval restaging:
  If restaging imaging positive will have Radical Neck Resection followed by Pembrolizumab 17 cycles, 200mg IV Q3W +/- External Beam Radiotherapy (if >10% viable tumour cells at resection) If restaging imaging negative will have Mapping biopsy. If biopsy positive will proceed to Radical Neck dissection followed by Pembrolizumab 17 cycles 200mg IV, Q3W If biopsy negative will proceed to Pembrolizumab 17 cycles 200mg IV, Q3W
  Interventions: Drug: Pembrolizumab

INTERVENTIONS:
Drug: Pembrolizumab — Delivery of neo-adjuvant Pembrolizumab
  Other Names: External Beam Radiation Therapy; Radical Neck Dissection

SUMMARY:
Cutaneous Squamous Cell Carcinoma (cSCC) is typically associated with a high tumour mutation burden, with the majority caused by Ultraviolet (UV) exposure (Pickering et al., 2014).

The use of this trial using neoadjuvant Pembrolizumab in patients with cSCC who will otherwise undergo highly morbid radical surgical resection has multiple potential advantages, including:

1. Reduction in surgical and radiotherapy morbidity by reducing tumour burden and allowing the appropriate selection of patients to undergo post-operative radiotherapy;
2. Provision of immediate information about pathological response and
3. Access to tissue to provide insight into resistance mechanisms and identification of biomarkers of response.

The Investigators hypothesized that the use of neoadjuvant Pembrolizumab could reduce tumour burden allowing appropriate selection of patients undergoing radical surgical resection and adjuvant radiotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed diagnosis of invasive cSCC that is locally advanced (Stage II-IV on AJCC 8th edition) assessed preoperatively as sufficiently high risk that they will warrant post-operatively RT (as recommended by MDT) who is a candidate for a complete resection.

Note: Participants with tumors arising on cutaneous non-glabrous (hair-bearing) lip with extension onto vermillion (dry red lip) may be eligible after communication and approval from the principal investigator. Participants for whom the primary site is the nose may be eligible after communication and approval from the MDT if the primary site is skin, not nasal mucosa with outward extension to skin. Participants who have squamous cell parotid metastases and have been treated previously for cSCC are permitted. cSCC that has recurred in the same location after 2 or more surgical procedures are not eligible.

* Participants must have measurable disease based on RECIST 1.1. Lesions situated in a previously irradiated area are considered measurable if progression has been demonstrated in such lesions.
* Participants must have an Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1 within 10 days prior to the start of treatment.
* Participants must have adequate organ function
* Participants must have a tissue sample adequate for translational research. This tissue sample may be obtained from either a newly obtained core or excisional biopsy.
* Participants must have a life expectancy of greater than 6 months.
* Be at least 18 years of age on the day of signing the informed consent. 8. Female participants: Female participants of childbearing potential must have a negative urine or serum pregnancy test within 72 hours prior to receiving the first dose of trial medication. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.

Note: In the event that 72 hours have elapsed between the screening pregnancy test and the first dose of study treatment, another pregnancy test (urine or serum) must be performed and must be negative in order for the participant to start receiving study medication.

- A female participant is eligible to participate if she is not pregnant, not breastfeeding, and at least one of the following conditions applies: Not a woman of childbearing potential (WOCBP) as defined in Appendix 1 OR A WOCBP who agrees to use an adequate method of contraception during the treatment period and for at least 120 days after the last dose of study treatment. Note: Abstinence is acceptable if this is the usual lifestyle and preferred contraception for the participant.

- The participant (or legally acceptable representative if applicable) must be willing and able to provide written informed consent for the trial. The participant may also provide consent for Future Biomedical Research. However the participant may participate in the main trial without participating in Future Biomedical Research.

Exclusion Criteria:

* Participant has metastatic/unresectable cSCC that cannot be potentially cured with surgical resection, radiotherapy, or with a combination of surgery and radiotherapy.
* Participant has any other histologic type of skin cancer other than invasive squamous cell carcinoma as the primary disease under study, eg, basal cell carcinoma that has not been definitively treated with surgery or radiation, Bowen's disease, merkel cell carcinoma, melanoma.
* Participants with any prior allogeneic solid organ or hematopoietic stem cell transplantations are excluded.
* Participant has received prior therapy with an anti-PD-1, anti-PD-L1, or anti-PD-L2 agent or with an agent directed to another stimulatory or co-inhibitory T-cell receptor (eg, CTLA-4, OX-40, CD137).
* Participant has received prior systemic anti-cancer therapy including investigational agents for cSCC.
* Participant has received prior radiotherapy to the target lesion.
* Participant has received a live vaccine within 30 days prior to the first dose of trial drug. Examples of live vaccines include, but are not limited to, the following: measles, mumps, rubella, varicella/zoster (chicken pox), yellow fever, rabies, Bacillus Calmette-Guérin (BCG), and typhoid vaccine. Seasonal influenza vaccines for injection are generally killed-virus vaccines and are allowed; however, intranasal influenza vaccines(eg, FluMist®) are live- attenuated vaccines and are not allowed.
* Participant is currently participating in or has participated in a trial of an investigational agent or has used an investigational device within 4 weeks prior to the first dose of trial treatment.

Note: Participants who have entered the follow-up phase of an investigational trial may participate as long as it has been 4 weeks after the last dose of the previous investigational agent.

* Ongoing or recent (within 2 years) evidence of significant autoimmune disease that required treatment with systemic immunosuppressive treatments, which may suggest risk for immune-related adverse events (irAEs) or has a diagnosis of immunodeficiency disorders (such as HIV disease or organ transplantation or hematologic malignancies associated with immune suppression).
* The following are not exclusionary: vitiligo; asthma; type 1 diabetes; hypothyroidism that required only hormone replacement; or psoriasis that does not require systemic treatment.
* Participant has a diagnosis of immunodeficiency or is receiving systemic steroid therapy (in dosing exceeding 10 mg daily of prednisone equivalent) or any other form of immunosuppressive therapy within 7 days prior the first dose of trial drug.
* Participant has a diagnosis and/or has been treated for additional malignancy within the past 3 years prior to allocation.

Note: Participants with cSCC of the skin that have undergone potentially curative therapy are not excluded if not related to current diagnosis.

Note: Participants with basal cell carcinoma of the skin or carcinoma in situ (eg, breast carcinoma, cervical cancer or melanoma in situ) that have undergone potentially curative therapy are not excluded.

Note: Participants with low-risk early-stage prostate cancer, defined as below are not excluded: Stage T1c or T2a with a Gleason score 6 and a prostate-specific antigen (PSA) (10 ng/ml) either treated with definitive intent or untreated in active surveillance that has been stable for the past year prior to trial allocation.

* Participant has an active autoimmune disease that has required systemic treatment in the past 2 years (eg, with use of disease-modifying agents, anticoagulants, corticosteroids or immunosuppressive drugs). Replacement therapy (eg, thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency) is not considered a form of systemic treatment and is allowed.
* Participant has a history of (non-infectious) pneumonitis that required steroids or has current pneumonitis.
* Participant has an active infection requiring systemic therapy.
* Participant has a known history of Hepatitis B (defined as Hepatitis B surface antigen [HBsAg] reactive) or known active Hepatitis C virus (defined as HCV RNA [qualitative] is detected) infection.

Note: No testing for Hepatitis B or Hepatitis C is required unless mandated by a local health authority.

* Participant has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the participant's participation for the full duration of the trial, or is not in the best interest of the participant to participate, in the opinion of the treating investigator.
* Participant has a known psychiatric or substance abuse disorder that would interfere with the participant's ability to cooperate with the requirements of the trial.
* Participant is pregnant or breastfeeding or expecting to conceive or father children within the projected duration of the trial, starting with the screening visit through 120 days after the last dose of trial treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Estimated)
Dates: Start 2022-06-28 (Actual); Primary Completion 2025-06-01 (Estimated); Study Completion 2027-06-01 (Estimated)

PRIMARY OUTCOMES:
Assess the rate of pathological response to neo-adjuvant Pembrolizumab | Will be assessed at the end of Cycle 4 (each cycle is 21 days) of Neo-adjuvant Pembrolizumab.
  To assess the rate of pathological response of neo-adjuvant Pembrolizumab in patients with locally advanced, resectable cSCC. Response will be measured by reviewing tissue samples taken at either surgical resection or biopsy following 4 cycles of neo-adjuvant Pembrolizumab. A pathological complete response will show no viable tumour cells.
  Pathological response will be determined as:
  Major Pathological response (less than or equal to 10% viable tumour cells remaining following 4 cycles of Neo-adjuvant Pembrolizumab) Pathological Partial Response (11-50% of viable tumour cells remaining following 4 cycles of neo-Adjuvant Pembrolizumab) Pathological Stable and/or Progressive disease (greater than 50% viable tumour cells following 4 cycles of Neo-adjuvant Pembrolizumab)

SECONDARY OUTCOMES:
Objective response Rate | Will be assessed at the end of Cycle 4 (each cycle is 21 days) of Neo-adjuvant Pembrolizumab
  To estimate objective response rate (ORR) as per investigator assessed RECIST 1.1 criteria
Disease free survival | From date of drug allocation until the date of first documented recurrence or date of death from any cause, whichever came first, assessed up to 48 months
  To estimate investigator assessed disease free survival (DFS) per RECIST 1.1 criteria
Overall Survival | From date of drug allocation until the date of death from any cause, whichever came first, assessed up to 48 months
  To evaluate the overall survival (OS) of the participants.
Locoregional Recurrence | From date of drug allocation until the date of first documented locoregional recurrence or date of death from any cause, whichever came first, assessed up to 48 months
  Freedom from locoregional recurrence
Distant Recurrence | From date of drug allocation until the date of first documented distant recurrence or date of death from any cause, whichever came first, assessed up to 48 months
  Freedom from Distant Recurrence
Incidence of Treatment Emergent Adverse Events related to Pembrolizumab | From date of study allocation until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 48 months
  Incidence of Treatment-Emergent Adverse Events as assessed by CTCAE Version 5
Number of Participants with Positive Surgical margins | At the end of Cycle 4 (cycle length 21 days)
  Positive surgical resection margin defined as tumour cells ≤5mm from the surgical margin.

OTHER OUTCOMES:
Rate of De-escalation of surgery or post-operative radiotherapy following neo-adjuvant pembrolizumab | At the end of 4 cycles of neo-adjuvant pembrolizumab. Each cycle is 21 days.
  Change from planned baseline multidisciplinary meeting recommendation. Patient may de-escalate both Post-operative radiotherapy +/- surgery depending on response
Pattern of failure | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 2 years following last administration of study drug (4 years total)
  Pattern of failure, assessed using descriptive analysis of percentages of patients in which disease recurrence for the primary endpoint of the study is due to local recurrence, regional recurrence, or distant recurrence
Cumulative occurrence of Second Primary Tumours (SPT) | From date of drug allocation until the date of first documented recurrence or date of death from any cause, whichever came first, assessed up to 48 months
  Cumulative occurrence of SPTs for each patient
18F FDG PET/CT complete metabolic response (CMR) rate | Assessed at the end of Cycle 4 (each cycle is 21 days)
  absence FDG uptake of target tumour lesion on 18F FDG PET/CT

CONTACTS AND LOCATIONS:
Overall Officials: Rahul Ladwa, MD, Principal Investigator — Queensland Health
Locations (3):
- Australia (3):
  - Chris O'Brien Lifehouse, Camperdown, New South Wales
  - Royal Brisbane and Women's Hospital, Herston, Queensland
  - Princess Alexandra Hospital, Woolloongabba, Queensland

IPD SHARING:
Plan to Share IPD: Yes
All individual data collected during trial in summary
Supporting Information: Study Protocol, CSR
Time Frame: Immediately following publication with no end date
Access Criteria: Available for sub-study, meta analysis

REFERENCES:
- [Derived] Ladwa R, Lee JH, McGrath M, Cooper C, Liu H, Bowman J, Gupta R, Cuscaden C, Nottage M, Clark JR, Le D, Pauley M, Kulasinghe A, Gonzalez-Cruz J, Porceddu SV, Hughes BGM, Panizza B. Response-Adapted Surgical and Radiotherapy De-Escalation in Resectable Cutaneous Squamous Cell Cancer Using Pembrolizumab: The De-Squamate Study. J Clin Oncol. 2025 Sep 10;43(26):2888-2896. doi: 10.1200/JCO-25-00387. Epub 2025 Jul 21. PMID 40690729